CLINICAL TRIAL: NCT01637181
Title: Comparative Randomized Clinical Trial of Endovenous 940 nm Laser Ablation Versus Endovenous 1470 nm Laser Ablation for Treatment of Great Saphenous Veins
Brief Title: Clinical Trial of Endovenous 940 and 1470 Laser Ablation for Treating Great Saphenous Veins
Acronym: COLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Wendy Malskat, MD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL38160.078.11
Record Dates: First submitted 2012-06-18; First posted 2012-07-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Varicose Veins; Insufficiency of Great Saphenous Vein
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- EVLA 940 nm (Active Comparator)
  Interventions: Procedure: Endovenous laser ablation (EVLA)
- EVLA 1470 nm (Active Comparator)
  Interventions: Procedure: Endovenous laser ablation (EVLA)

INTERVENTIONS:
Procedure: Endovenous laser ablation (EVLA) — EVLA with 940 nm Diode laser EVLA with 1470 nm Nd:Yag laser With both devices, obliteration of the varicose vein is obtained by heating the vein, using emission of laser light.

SUMMARY:
A clinical randomized controlled trial, comparing 2 endovenous laser ablation (EVLA) techniques in patients with insufficiency of the great saphenous vein (GSV). There are multiple EVLA devices available, with different wavelengths. In the Netherlands, 940 nm Diode and 1470 nm Nd:Yag laser are the most frequently used devices. Both devices also proven to be equally effective in occluding the GSV. However, little is known about differences in patient-related outcomes. Therefore, the primary outcomes of this comparative clinical trial of 940 nm and 1470 nm EVLA, are pain scores, patient satisfaction and scores of health related and varicose-specific questionnaires. The secondary outcomes are complications and effectiveness of the treatment. It is thought that possibly the 1470 nm ELVA will give lower pain scores and higher patient satisfaction than 940 nm EVLA. No differences are expected in complication rate and effectiveness between the two treatments.

DETAILED DESCRIPTION:
* Study type: Interventional. Randomized comparative clinical trial..

* Outcome measures:

  * Primary study outcomes: Patient reported outcomes: 1. Pain score and use of painkillers, assessed with a numeric rating scale (NRS) of pain. 2. Treatment satisfaction, assessed with a NRS of satisfaction. 3. Health related quality of life, assessed with Dutch translated Aberdeen Varicose Vein Questionnaire (AVVQ) and EQ-5D questionnaire.
  * Secondary study outcomes: 1. Number of patients with adverse events. Major complications: deep and superficial venous thrombosis (embolic events), nerve injury, skin burns, and (sub)cutaneous infections. Minor complications: ecchymosis and hyperpigmentation. 2. Obliteration of varicose vein and/or absence of reflux (> 0.5 sec. of retrograde flow) along the treated segment of the GSV. This is measured using US examination.
* Outcome measures time frame:

Follow-up of one year, with outcome measures at baseline, 1 week, 3 months and 1 year post treatment.

* Focus of the study: Varicose great saphenous veins (GSV)

* Intervention information:

  * Intervention name: endovenous laser ablation (EVLA)
  * Intervention type: 1. EVLA with 940 nm Diode laser 2. EVLA with 1470 nm Nd:Yag laser
  * Arm information: both interventions are active comparators.
* Locations:

Rotterdam, Zuid-Holland, The Netherlands

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Insufficiency of the GSV measured with ultrasound imaging, reflux > 0.5 sec, and diameter of vein > 0.5 cm
* Symptoms of chronic venous insufficiency, including complaints related to varicose veins (≥ C2)
* No prior treatment of the insufficient GSV
* Informed consent

Exclusion Criteria:

* Acute deep or superficial vein thrombosis
* Agenesis of deep vein system
* Vascular malformation or syndrome
* Post-thrombotic syndrome, occlusive type
* Pregnancy
* Immobility
* Allergy to lidocaine
* Arterial insufficiency
* Diameter of GSV ≤ 0.5 mm at puncture site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain score and use of painkillers | 1 week post treatment
  A questionnaire including a numeric rating scale (NRS) of pain is filled in by the patient.
Treatment satisfaction | 1 week post treatment
  A NRS of satisfaction is filled in by the patient.
Health related quality of life | 0 and 12 weeks post treatment
  Dutch Translated Aberdeen Varicose Vein Questionnaire (AVVQ) and EQ-5D questionnaire are filled in by the patient.

SECONDARY OUTCOMES:
Number of participants with adverse events | The adverse events will be assessed at 1 and 12 weeks post treatment.
  Minor complications: ecchymoses and hyperpigmentation. Major complications: deep and superficial venous thrombosis (embolic events), nerve injury, skin burns, and (sub)cutaneous infections.
Occlusion of the treated GSV (effectiveness) | The rates will be compared between 940 nm and 1470 nm endovenous laser at time 1, 12 and 52 weeks post treatment.
  Obliteration of varicose vein and/or absence of reflux (>0.5 sec. of retrograde flow) along the treated segment of the GSV. This is measured using US examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

REFERENCES:
- [Derived] Malskat WS, Giang J, De Maeseneer MG, Nijsten TE, van den Bos RR. Randomized clinical trial of 940- versus 1470-nm endovenous laser ablation for great saphenous vein incompetence. Br J Surg. 2016 Feb;103(3):192-8. doi: 10.1002/bjs.10035. Epub 2015 Dec 14. PMID 26661521